CLINICAL TRIAL: NCT07340164
Title: A Phase 2, Open-label, Multicenter, Randomized Study of Trastuzumab Deruxtecan Versus Investigator's Choice Chemotherapy in Recurrent Ovarian Cancer That Progressed on Prior PARP Inhibitor Therapy: TROY (APGOT-OV14)
Brief Title: Trastzumab Deruxtecan Versus SOC in Recurrent Ovarian That Progressed on Prior PARP Inhibitor Therapy
Acronym: TROY
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Daiichi Sankyo (Industry); Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, JUNGYUN LEE, professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2025-1110
Record Dates: First submitted 2025-12-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma, Recurrent; Ovarian Cancer Metastatic Recurrent; Ovarian Cancer (OvCa)
Keywords: TROY; APGOT-OV14; ENGOT-ov92
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — trastuzumab deruxtecan; Bevacizumab; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Trastzumab Deruxtecan(T-DXd) +/- Bevacizumab
  Interventions: Drug: Trastzumab Deruxtecan; Drug: Bevacizumab
- Arm B (Active Comparator): Platinum based chemotherapy +/- Bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Platinum Based Chemotherapy

INTERVENTIONS:
Drug: Trastzumab Deruxtecan — Trastzumab deruxtecan will be administrated via intravenous, every 3 weeks.
  Other Names: T-DXd; Enhertu; DS-8201
  Arms: Arm A
Drug: Bevacizumab — Bevacizumab is administered intravenously in one of two doses: 1. 10 mg/kg every 2 weeks 2. 15 mg/kg every 3 weeks
  1. 10mg/kg, every 2weeks
  2. 15mg/kg, every 3weeks
Drug: Platinum Based Chemotherapy — *Proposed regimens for Arm B
  1. PLD 30~40mg/m2 D1 + Carboplatin AUC 5 D1 +/- bevacizumab 10mg/kg D1/D15 q4w (for 6-8 cycles) followed by bevacizumab 15mg/kg q3w
  2. Paclitaxel 175mg/m2 D1 + Carboplatin AUC 5 D1 +/- bevacizumab 15mg/kg D1 q3w (for 6-8 cycles) followed by bevacizumab 15mg/kg q3w
  3. Gemcitabine 1000mg/m2 D1/D8 + Carboplatin AUC 4 or 5 D1 +/- bevacizumab 15mg/kg D1 q3w (for 6-8 cycles) followed by bevacizumab 15mg/kg q3w
  Arms: Arm B

SUMMARY:
Ovarian, fallopian tube, and peritoneal cancers are often diagnosed at an advanced stage, requiring chemotherapy. Recently, the standard treatment, platinum-based chemotherapy plus PARP inhibitors, has extended disease-free survival (PFS). However, most patients eventually develop resistance to PARP inhibitors and become unresponsive to conventional treatments. Therefore, an effective standard treatment for patients who relapse after PARP inhibitor resistance has not yet been established. Meanwhile, HER2 protein expression has been identified in some patients, drawing attention as a new therapeutic target.

Trastuzumab deruxtecan (T-DXd), an antibody-drug conjugate (ADC) targeting HER2, has already demonstrated efficacy and safety in other HER2-positive cancers. This study aimed to explore the potential of T-DXd as a new treatment option by evaluating the efficacy and safety of T-DXd in patients with ovarian, fallopian tube, and peritoneal cancer who relapsed after PARP inhibitor treatment and who express HER2.

Participants will:

* Arm A: T-DXd +/- Bevacizumab, IV, every 3weeks
* Arm B: Platinum-based chemotherapy +/- Bevacizumab, IV

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults ≥18 years of age on the day of signing the Informed Consent Form. Follow local regulatory requirements if the legal age of consent for trial participation is >18 years old.

  2. Patient has signed the Informed Consent (ICF) and is able to comply with protocol requirements.

  3. Has HER2 expression per 2016 ASCO-CAP gastric cancer IHC scoring (3+/2+/1+) guidelines by local tests.

  4. Availability of tumor tissue for translational research: A formalin-fixed paraffin-embedded (FFPE) tumorblock (preferred) or at least 20 slides (unstained, freshly cut, serial sections) must be submitted.

  5. Histologically confirmed high grade serous or high grade endometrioid ovarian, primary peritoneal, and/or fallopian tube cancer that is recurrent.

  6. Patient with an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

  7. Radiologically confirmed/documented disease progression while on PARP inhibitor therapy in either first or second-line maintenance setting Note: Documentation of disease progression must be within 180 days of last PARPi dose taken. Surgical salvage intervention and/or focal ablative therapies are allowed.
  1. Clinically benefited from PARPi maintenance prior to documented progression, as defined by at least 6 months of treatment duration with no progressive disease observed.
  2. Progression on first-line maintenance PARP inhibitor: Participants are allowed maximum 1 additional line of platinum-based chemotherapy before study entry (note: treatment-free interval on platinum rechallenge must be > 6 months, with documented disease progression prior to study entry.
  3. Progression on second-line maintenance PARP inhibitor: Participants are not allowed any additional systemic anticancer treatment before study entry.

     8. Patient with measurable disease according RECIST 1.1 criteria. 9. LVEF ≥50% within 28 days before randomization. 10. Patient has adequate organ function, defined as follows:

  a) Absolute neutrophil count ≥ 1,500 cells/μL b) Platelets ≥ 100,000 cells/μL c) Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L d) Serum creatinine ≤ 1.5× upper limit of normal (ULN) or calculated creatinine clearance ≥ 50mL/min using the Cockcroft-Gault equation for patients with creatinine levels > 1.5× institutional ULN e) Total bilirubin ≤ 1.5× ULN (≤ 2.0 x ULN in patients with known Gilbert's syndrome) or direct bilirubin ≤ 1× ULN f) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN unless liver metastases are present, in which case they must be ≤ 5× ULN g) International normalized ratio or prothrombin time (PT) ≤1.5× ULN and activated partial thromboplastin time ≤1.5× ULN. Patients receiving anticoagulant therapy must have a PT or partial thromboplastin within the therapeutic range of intended use of anticoagulants.

  11. Patient must have a negative serum pregnancy test within 72 hours of the first dose of study medication, unless they are of nonchildbearing potential. Nonchildbearing potential is defined as follows:
  1. Patient is ≥ 45 years of age and has not had menses for > 1 year.
  2. A follicle-stimulating hormone value in the postmenopausal range upon screening evaluation if amenorrhoeic for < 2 years without a hysterectomy and oophorectomy.
  3. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation:
* Documented hysterectomy or bilateral oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound, MRI, or CT scan.
* Tubal ligation must be confirmed with medical records of the actual procedure.
* Information must be captured appropriately within the site's source documents. 12. Patient of childbearing potential must agree to use a highly effective method of contraception with their partners starting from time of consent through 150 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient (Information must be captured appropriately within the site's source documents) 13. Has proteinuria <2+. If proteinuria is ≥2+, 24-hour urine must demonstrate <1 g of protein in 24 hours.

Exclusion Criteria:

- 1. Primary platinum-refractory disease defined as disease progression during primary platinum-based chemotherapy or platinum-resistant disease defined as disease progression within 6 months of the last platinum administration in the second-line setting.

2. History of additional malignancy within 3 years before the date of enrolment. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, with concurrence of the Sponsor, is considered cured with minimal risk of recurrence within 3 years. 3. Patient has received prior anticancer therapy (chemotherapy, targeted therapies, hormonal therapy, radiotherapy) within 21 days or < 5 times the half-life of the most recent therapy prior to Study Day 1, whichever is shorter.

Note: The washout period for radiation therapy is as follows: ≥ 4 weeks for palliative stereotactic radiation to chest and ≥2 weeks palliative stereotactic radiation therapy to other anatomic areas.

4. Patient has known uncontrolled central nervous system metastases, carcinomatosis meningitis, or both.

Note: Patients with previously treated brain metastases may participate provided they are stable (without evidence of disease progression by imaging [using the identical imaging modality for each assessment, either MRI or CT scan] for at least 4 weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and have not been using steroids for at least 7 days prior to study treatment. Carcinomatous meningitis precludes a patient from study participation regardless of clinical stability. 5. Active and/or uncontrolled infection. The following exceptions apply:

1. Participants with HIV infection are eligible if followings are met: a. CD4+ T-cell count ≥350 cells/mm3 at the time of screening, b. Virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) at the time of screening and for at least 12 weeks before screening, c. No AIDS-defining opportunistic infections or conditions within the past 12 months, d. On stable ART regimen, without changes in drugs or dose modification, for at least 4 weeks before trial entry (Day 1) and agree to continue ART throughout the trial.
2. Participants with evidence of chronic HBV infection are eligible if the followings are met: a. the HBV viral load is <2000 IU/mL b. start or maintain antiviral treatment, if clinically indicated as per the investigator. c. they have normal transaminase values, or, if liver metastases are present, abnormal transaminases with a result of AST/ALT <3 × ULN, which are not attributable to HBV infection.
3. Participants with a history of HCV infection are eligible if History of hepatitis C infection eligible if the HCV viral load is below the level of detection in the absence of antiviral therapy during the previous 4 weeks and if they Have normal transaminase values, or, if liver metastases are present, abnormal transaminases with a result of AST/ALT <3 × ULN, which are not attributable to HCV infection.

   6. Patient has not recovered (i.e., to Grade ≤ 1 or to baseline) from cytotoxic therapy-induced adverse events(AEs).

Note: Patients with Grade ≤ 2 neuropathy, Grade ≤ 2 alopecia, or Grade ≤ 2 fatigue are an exception to this criterion and may qualify for the study.

7. Patient has not recovered adequately from AEs or complications from any major surgery prior to starting therapy.

8. Patient has a known hypersensitivity to the active substances or to any excipients of the study intervention 9. Evidence of active or ongoing bowel obstruction 10. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.

11. Uncontrolled or significant cardiovascular disease, including the following:

1. QT interval corrected with Fridericia's formula interval >470 ms (average of triplicate determinations).
2. Diagnosed or suspected long QT syndrome or known family history of long QT syndrome.
3. History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes.
4. Myocardial infarction within 6 months prior to screening.
5. Uncontrolled angina pectoris within 6 months prior to screening.
6. New York Heart Association Class 2 to 4 congestive heart failure.
7. Patients with uncontrolled hypertension (defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥100 mmHg) based on an average of ≥ 3 BP readings on ≥ 2 sessions.
8. Complete left or right bundle branch block.
9. Patients with troponin levels above ULN at screening (as defined by the manufaccturer), and wit any MI related symptoms. (For patients with elevated troponin levels but no MI symptoms, a cardiology consultation during the screening period is recommended..

   12. Patient is currently participating and receiving study treatment or has participated in a study of an investigational agent and received study treatment or used an investigational device within 4 weeks of the first dose of treatment.

   13. Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation) 14. Patients with current abdominal/ pelvic fistula. 15. Patient is considered a poor medical condition due to a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active infection requiring systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled ventricular arrhythmia; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study(including obtaining informed consent).

   16. Prior exposure to other HER2-targeted agents or antibody-drug conjugate that consists of an exatecan derivative that is a topoisomerase I inhibitor 17. Patient is pregnant or breastfeeding or is expecting to conceive children within the projected duration of the study, starting with the screening visit through 7 months after the last dose of study treatment, or lactating woman.

   18. Live vaccines within 30 days of first dose of study intervention and while receiving study intervention. Administration of inactivated vaccines (i.e. inactivated influenza vaccine) is permitted. Inactivated RNA or nonreplicating viral vector-based SARS-CoV-2 vaccines are allowed, as approved by local/regional Health Authorities. Novel live attenuated SARS-CoV-2 vaccines are not permitted.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in HER2 IHC 1+/2+/3+ population | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Defined as the time from the date of randomization until first documentation of disease progression, as determined by investigator assessment based on RECIST 1.1, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) in HER2 IHC 2+/3+ population | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Defined as the time from the date of randomization until first documentation of disease progression, as determined by investigator assessment based on RECIST 1.1, or death due to any cause, whichever occurs first
Objective Response Rate (ORR) by investigator in HER2 2+/3+ population | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Defined as the proportion of patients who have best overall response of either complete response (CR) or partial response (PR), as investigator assessment based on RECIST 1.1
Objective Response Rate (ORR) by investigator in HER2 1+/2+/3+ population | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Defined as the proportion of patients who have best overall response of either complete response (CR) or partial response (PR), as investigator assessment based on RECIST 1.1
Disease control rate (DCR) by investigator in HER2 2+/3+ population | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Defined as the proportion of patients who have best overall response of CR, PR, or stable disease (SD) by investigator assessment per RECIST 1.1 . SD must be achieved at ≥ 7 weeks after randomization to be considered best overall response.
Disease control rate (DCR) by investigator in HER2 1+/2+/3+ population | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Defined as the proportion of patients who have best overall response of CR, PR, or stable disease (SD) by investigator assessment per RECIST 1.1 . SD must be achieved at ≥ 7 weeks after randomization to be considered best overall response.
Clinical benefit rate (CBR) by investigator in HER2 2+/3+ population | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Defined as the proportion of patients who have best overall response of CR, PR, or stable disease (SD) by investigator assessment per RECIST 1.1 . (duration of SD ≥ 23 weeks after randomization)
Clinical benefit rate (CBR) by investigator in HER2 1+/2+/3+ population | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  Defined as the proportion of patients who have best overall response of CR, PR, or stable disease (SD) by investigator assessment per RECIST 1.1 . (duration of SD ≥ 23 weeks after randomization)
Duration of Response Rate (DoR) by investigator in HER2 2+/3+ population | From the time of first documentation of CR or PR until the time of first documentation of subsequent PD or death from any cause, whichever came first, assessed up to 5 years.
  Measured from the time of initial response until documented tumor progression.
Duration of Response Rate (DoR) by investigator in HER2 1+/2+/3+ population | From the time of first documentation of CR or PR until the time of first documentation of subsequent PD or death from any cause, whichever came first, assessed up to 5 years.
  Measured from the time of initial response until documented tumor progression.
Time to first subsequent treatment (TFST) Time to second Subsequent Treatment (TSST) in HER2 2+/3+ population | From the date of randomization to date of the first and second subsequent anticancer therapy or death, whichever came first, assessed up to 5 years.
  Defined as the time from the date of randomization to date of the first and second subsequent anticancer therapy or death.
Time to first subsequent treatment (TFST) Time to second Subsequent Treatment (TSST) in HER2 1+/2+/3+ population | From the date of randomization to date of the first and second subsequent anticancer therapy or death, whichever came first, assessed up to 5 years.
  Defined as the time from the date of randomization to date of the first and second subsequent anticancer therapy or death.
Progression free survival 2 (PFS2) measured by investigator in HER2 1+/2+/3+ population | the time from treatment randomization to the earlier date of assessment of progression on the next anticancer therapy following study treatment or death by any cause, whichever came first, assessed up to 5 years.
  Defined by the time from initial randomization to the second objective disease progression (ie, after the first subsequent therapy) or death.
OS in the HER2 IHC 2+/3+ population | the time from the date of inclusion until death due to any cause, assessed up to 5 years.
  Measured as the time from the date of randomization to the date of death
OS in the HER2 IHC 1+/2+/3+ population | the time from the date of inclusion until death due to any cause, assessed up to 5 years.
  Measured as the time from the date of randomization to the date of death
Response rate of subsequent therapies | From the start date of subsequent anticancer therapy until death due to any cause or study termination, assessed up to 5 years.
  Defined as the proportion of patients who have best overall response of either complete response (CR) or partial response (PR), as investigator assessment based on RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No